CLINICAL TRIAL: NCT03301922
Title: Metacognitive Therapy and Work Interventions for Patients on Sick Leave Due to Common Mental Disorders: A Randomized Waiting List Controlled Trial
Brief Title: Metacognitive Therapy and Work Interventions for Patients on Sick Leave Due to Common Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1794
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Anxiety; Depression
Keywords: Occupational Health Services; Metacognitive therapy; Work focused interventions; Sick leave
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Work-focused metacognitive therapy (Experimental): Work-focused metacognitive therapy
  Interventions: Behavioral: Metacognitive therapy and work-focused interventions
- Waiting list (Other): Waiting list
  Interventions: Behavioral: Metacognitive therapy and work-focused interventions; Other: Waiting list

INTERVENTIONS:
Behavioral: Metacognitive therapy and work-focused interventions — Metacognitive therapy and work-focused interventions, up to maximum 12 sessions, with weekly session of 45-60 minute duration. The metacognitive treatment program is based on Wells' manual. The work-focused intervention is based on Lagerveld and Blonk. The interventions are run in parallel.
Other: Waiting list — Waiting list
  Arms: Waiting list

SUMMARY:
Common mental health disorders such as anxiety and depression are leading causes of sickness absence and disability in Norway. Despite tremendous costs for individual and society, effective treatment is lacking. Mental health interventions do not typically target work situation, despite its importance for patient well-being. On a policy level, effective measures are impeded by a paucity of scientific data, and programs designed to address the issue such as Faster Return to Work ("Raskere tilbake") lack evaluation. The present project will test the effectiveness of Metacognitive therapy and work-focused interventions for reducing sick leave in patients with common mental disorders.

DETAILED DESCRIPTION:
Common mental health disorders (CMD) such as anxiety and depression are leading contributors to the global burden of disease , generating substantial costs for societies in reduced productivity and increased benefit pay outs. In 2010, the worldwide cost of mental health disability was estimated at US$2.5-8.5 trillion in lost output, and the sum is projected to double by 2030 unless effective policy measures are implemented. For middle- and high-income countries, 30-50 % of disability applications stem from mental health issues, and the proportion is likely greater among the younger part of the work force. In Europe, depression is responsible for 13.7 % of all years lived with disability, and anxiety disorders likely have similar impact. Mental health issues are among the leading causes of disability and early retirement across the European region.

For affected individuals, anxiety and depression reduces quality of life, decreases functioning and increases the risk of further health problems. Sick leave is often used for adults with CMD, but may not always be helpful. Avoidance and isolation are behavioural strategies that maintain anxiety and depression. Absenteeism from work, an important social arena, may strengthen this behaviour, impeding recovery. Even when controlling for the impact of ill health, short term sick leave may in itself increase the risk of future long term absence. In addition, employment rates are 10-15% lower for people with mental ill health than the rest of the population. Exclusion from the work force is in turn associated with poorer mental health, and can heighten the risk of futures depression and even suicide. The relationship between CMD and reduced work-participation is therefore likely bidirectional, and sick leave may not work as intended despite its high cost for society.

The individual and societal burden from sick leave and mental health represents a key policy challenge on the global agenda and the need for efficient measures is urgent. Norway exemplifies this urgent need as expenditure on disability and sickness absence totals 5 % of GDP, by far the highest in the OECD. Efforts have been made to address the issue through several policy initiatives, such as the nationwide Faster Return to Work (FRW) program. The program facilitates buying treatment from different actors to reduce waiting times and thus potentially the duration of sick leave. The impact of the program is uncertain, as little research has been done on its efficacy. Scientific data on Norwegian sick leave follow up is mostly absent. Despite the magnitude of the challenge, there is a clear knowledge gap.

Investment in sick leave follow up has not been equally distributed amongst patient groups. Sixty per cent of all working days lost to disability or sick leave are due to mental health issues and musculoskeletal complaints. Sick leave due to CMD is growing. When caused by mental health issues, disability pension is awarded on average nine years earlier than for somatic reasons, resulting in more working years lost to disability. Though prevalent in the statistics, few CMD patients on sick leave receive treatment. Only 1.4 % of employees on sick leave are referred to specialized mental health treatment. As many as one in three people awarded disability pension for mental illness have never received any form of treatment prior to disability being granted. This shows a severe under-referral and under-treatment for this patient group despite being responsible for the majority of sick leave and disability costs.

A more targeted approach, integrating work-focused interventions with effective CMD treatment is needed for this patient group. Two recent studies have examined such an approach. In the Netherlands, Lagerveld and Blonk conducted a randomized controlled trial where 168 patients on sick leave due to CMD received either cognitive behavioural therapy (CBT), or CBT with an integrated work-focused intervention. Their results showed a 20 % decrease in sickness absence for patients receiving the work-focused intervention, while maintaining effective symptom reduction. In Germany, similar results were found with a smaller sample size. A multicentre trial in Norway looked at registry data for 1193 CMD patients receiving a variation of work-specific interventions, showing a clear reduction in sick leave and disability. Integrated work-focused treatment for CMD is thus a promising avenue of research.

Metacognitive therapy (MCT) is a treatment based on more recent theoretical developments. It has shown excellent results for anxiety and depression, and the treatment protocol for generalized anxiety disorder and social phobia is recommended in the NICE guidelines. Rather than challenging and changing specific thought content (CBT), metacognitive treatment aims to change and challenge maladaptive cognitive processes, among these rumination and worry, which are key components in CMD and sick leave.

The study will be a randomized controlled trial. Participants will be persons with a primary diagnosis of common mental disorders, anxiety and depression. Experienced independent diagnosticians will assess all patients by using structural interviews MINI (MINI International Neuropsychiatric Interview).

All patients will be randomized in blocks to two groups in order to compare the following conditions: MCT and work-focused interventions, and a wait list control condition. After the waiting period of either 8 or 12 weeks, the patients in the wait-list condition will be allocated to the treatment condition. Both between-subjects and within-subjects comparisons will be conducted.

Questions that will be addressed are:

1. MCT and work-focused interventions will be superior to the wait-list condition in make participants return to work
2. Which changes in predictors related to treatment predict return to work
3. MCT and work-focused interventions will be superior to the wait-list condition for improving mental health
4. MCT and work-focused interventions will be more cost-efficient than the wait-list condition
5. Evaluate the sustainability of return to work for patients on sick leave due to common mental disorders after MCT and work-focused interventions
6. Examine impact of different potential prognostic factors on work function, both at the end of treatment and at one year follow-up.
7. If the effect of MCT and work-focused interventions will sustain one year after the end of therapy
8. Explore if patients will have reduced use of sick leave in the four years following after treatment compared to the two years prior to treatment based on register data.

The meta-cognitive treatment program is based on Wells' manual. The work-focused intervention is based on an adopted Norwegian version of Lagerveld and Blonk. The interventions are run in parallel. The patients who are receiving MCT and work-focused interventions will be treated up to maximum 12 sessions, with weekly session of 45-60 minute duration.

The treatment will be administered according to the originators published treatment protocols for MCT.

1. All patients referred to the clinic will be consecutively assessed at intake (MINI). Based on diagnosis and criteria for inclusion and exclusion, the patients will be asked to volunteer to participate in the study and confirm by signing a form of consent.
2. Patients will be randomized to one of the two conditions.
3. Patients will be asked to self-rate symptoms on a battery of self-report questionnaires.
4. Work-focused meta-cognitive therapy will be given to patients in group 1, while group 2 is a waiting list control. Waiting list controls will be rated but not treated and will wait for treatment for either 8 or 12 weeks.
5. After waiting they will be transferred to the treatment group.
6. The patients will be assessed prior to treatment, by at end of treatment weeks in treatment, and at six months and at, one and two years of follow-up.
7. Reassessment of the diagnosis and symptom severity is made by post-treatment.

Criteria for recovery will be: Jacobsen criteria of a minimum change and patients crossing the cut-off point on two measures: The BDI and BAI. Other outcome measures will include:

* Reduction of depressive symptoms as measured by self-report questionnaires
* Number of patients with no diagnosis based on MINI after treatment
* Relapse rate during six months and at, one year follow-up

A comparison between the two groups of patients will be conducted at post-treatment. Follow-up data will be analysed based on 6 month and at one year of follow up for the treatment condition with self-report and a four year follow-up with register data. A within group analyses will be conducted in order to estimate effect sizes and significant clinical change estimates.

Participants will be randomized in patients divided on three conditions in a 1:2 ratio. One factors are controlled for in the randomization, namely, gender. A computer program provided by NTNU WebCRF will generate the randomization list.

ELIGIBILITY:
Inclusion Criteria:

* on sick leave either partial or full, due to
* clinically relevant level of anxiety and depression, and
* eligible for work-related sick leave pay outs
* given consent

Exclusion Criteria:

* Serious mental illness (such as bipolar disorder or schizophrenia)
* Substance abuse
* Cluster A and B personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Changes in degree of sick leave | From 2 years prior to intervention - to 4 years after intervention
  data from National registers
Changes in degree of sick leave | From 2 years prior to intervention - to 4 years after intervention
  data from patients self-report
Changes in anxiety symptoms | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes in depressive symptoms measured by Beck Anxiety Inventory (BAI)
Changes in depressive symptoms | From pre treatment, to post treatment (12 weeks), 6 months 1 year follow-up
  Changes in depressive symptoms measured by Beck Depression Inventory II (BDI-II)

SECONDARY OUTCOMES:
Changes in metacognitions | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes in metacognitions symptoms measured by the Metacognitions Questionnaire 30 (MCQ-30)
Changes in subjective health complaints | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes in symptoms measured by Subjective Health Complaints
Changes in bullying and victimisation at work | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes in measured Negative Acts Questionnaire
Changes in self-efficacy | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes measured with Return to work self-efficacy
Changes in resilience | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes measured with The resilience scale for adults (RSA)
Changes in quality of life | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Changes measured with EQ-5D-5L
MINI - diagnostic interview | From pre treatment, to post treatment (12 weeks)
  Diagnostic evaluations using MINI - International Neuropsychiatric Interview

OTHER OUTCOMES:
Secondary analysis related to the onset of Covid-19 | From pre treatment, to post treatment (12 weeks), 6 months and 1 year follow-up
  Sub-analyses taking into consideration the onset of Covid-19 in Norway by mid March 2020

CONTACTS AND LOCATIONS:
Overall Officials: Odin Hjemdal, prof, Principal Investigator — Norwegian University of Science and Technology; Ragne GH Gjengedal, Study Chair — Diakonhjemmet Hospital
Locations (1):
- Poliklinikken Raskere Tilbake, Diakonhjemmet Sykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gjengedal RGH, Hannisdal M, Osnes K, Reme SE, Wells A, Blonk R, Lending HD, Johnson SU, Lagerveld SE, Anyan F, Nordahl HM, Gerritsen RBTW, Bjorndal MT, Wright D, Sandin K, Bjontegard KS, Schwach J, Hjemdal O. Metacognitive therapy and work-focus for patients with depression, anxiety or comorbid depression and anxiety on sick leave: a single-centre, open-label randomised controlled trial. EClinicalMedicine. 2025 Nov 6;89:103613. doi: 10.1016/j.eclinm.2025.103613. eCollection 2025 Nov. PMID 41357335
- [Derived] Sandin K, Gjengedal RGH, Osnes K, Hannisdal M, Berge T, Leversen JSR, Rov LG, Reme SE, Lagerveld S, Blonk R, Nordahl HM, Shields G, Wells A, Hjemdal O. Metacognitive therapy and work-focused interventions for patients on sick leave due to anxiety and depression: study protocol for a randomised controlled wait-list trial. Trials. 2021 Nov 27;22(1):854. doi: 10.1186/s13063-021-05822-4. PMID 34838125